CLINICAL TRIAL: NCT02685397
Title: The Role of Stereotactic Body Radiotherapy in the Management of Castration-Resistant Prostate Cancer with Oligometastases: an Adaptive Phase II/III Randomized Trial.
Brief Title: Management of Castration-Resistant Prostate Cancer with Oligometastases
Acronym: PCS IX
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Tamim Niazi, Principal Investigator, Sir Mortimer B. Davis - Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS IX
Record Dates: First submitted 2016-02-03; First posted 2016-02-18 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Castration-resistant Prostate Cancer Patients with Oligometastases
MeSH Terms: interventions — Leuprolide; luprolide acetate gel depot; Goserelin; Triptorelin Pamoate; enzalutamide; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

ARMS (2):
- LHRH agonist + Enzalutamide (Active Comparator): Subjects will receive LHRH agonist in combination with the new generation of hormonal therapy (enzalutamide, 40mg)
  Interventions: Drug: Leuprolide Acetate; Drug: Goserelin Acetate; Drug: Triptorelin; Drug: Enzalutamide
- LHRH agonist + Enzalutamide + SBRT (Experimental): Subjects will receive LHRH agonist in combination with the new generation of hormone therapy (enzalutamide, 40mg) plus the additional SBRT treatment
  Interventions: Drug: Leuprolide Acetate; Drug: Goserelin Acetate; Drug: Triptorelin; Drug: Enzalutamide; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Leuprolide Acetate — Luteinizing hormone releasing hormone (LHRH) agonist administered by subcutaneous injection. Only one of the LHRH agonists described here will be administered during the course of treatment.
  Other Names: Eligard; Lupron
Drug: Goserelin Acetate — Luteinizing hormone releasing hormone (LHRH) agonist administered by subcutaneous injection. Only one of the LHRH agonists described here will be administered during the course of treatment.
  Other Names: ZOLADEX
Drug: Triptorelin — Luteinizing hormone releasing hormone (LHRH) agonist administered by subcutaneous injection. Only one of the LHRH agonists described here will be administered during the course of treatment.
  Other Names: Trelstar
Drug: Enzalutamide — Anti-androgen medication for the treatment of metastatic castration-resistant prostate cancer. 160 mg (four 40 mg capsules) taken as a single oral daily dose, with or without food, until disease progression.
  Other Names: Xtandi
Radiation: Stereotactic Body Radiation Therapy — Stereotactic body radiation therapy (SBRT) is a treatment modality in radiation oncology that delivers a very high dose of radiation to the tumour target with high precision using a single or a small number of fractions.
  Other Names: SBRT
  Arms: LHRH agonist + Enzalutamide + SBRT

SUMMARY:
This adaptive phase II/III randomized trial is designed to demonstrate that eradication of oligometastases by SBRT is a promising and emerging way to delay disease progression and postpone second line systemic therapies in castration-resistant prostate cancer (CRPC) patients. Only CRPC patients with an oligometastatic recurrence will be eligible to take part in this trial. All participating patients will receive either the standard of care (i.e. LHRH agonist in combination with the new generation of hormonal therapy [Enzalutamide]) or the experimental treatment (i.e. LHRH agonist in combination with the new generation of HT [Enzalutamide] plus the additional SBRT treatment). The patients will undergo different evaluations before treatment, such as imaging to confirm oligometastatic recurrence and blood tests. Patients will be stratified according to the location of metastasis (visceral [with or without bone metastases] vs. bone metastases alone) and PSA doubling time (≤ 3 vs. > 3 months). As per the standard of care, patients will have PSA testing performed every 6-12 weeks and re-imaging at 6, 9, 12, 18 and 24 months or at PSA progression, whichever occurs first.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most common type of cancer to affect men and, unfortunately, for the majority of PCa patients, death is attributed to metastatic disease. Lifelong androgen deprivation therapy (ADT) with LHRH agonists can help delay cancer progression in metastatic PCa patients. However, patients eventually become castration-resistant (disease progression despite ADT) and develop progressive metastatic disease. This in turn impacts the patient's quality of life and survival. Recently, a new generation of hormonal therapy (such as Enzalutamide) has become available to these castration-resistant prostate cancer (CRPC) patients. We believe that the benefits from this new generation of hormonal therapy can be prolonged in CRPC patients who develop oligometastases by treating the metastatic lesions using stereotactic body radiotherapy (SBRT). This new radiation technique allows for the treatment of many different metastases throughout the body in a very precise manner. This metastases-directed therapy is a new treatment option for patients with a limited number of metastases (less than 5) at the time of recurrence.

This adaptive phase II/III randomized trial is designed to demonstrate that eradication of oligometastases by the new technique SBRT is a promising and emerging way to delay disease progression and to postpone second line systemic therapies. Only patients with an oligometastatic recurrence after local treatment with curative intent will be eligible to take part in this trial. All participating CRPC patients with oligometastases will receive either the standard of care (i.e. LHRH agonist in combination with the new generation of hormonal therapy [Enzalutamide]) or the experimental treatment (i.e. LHRH agonist in combination with the new generation of HT [Enzalutamide] plus the additional SBRT treatment). The patients will undergo different evaluations before treatment, such as imaging to confirm oligometastatic recurrence and blood tests. Patients will be stratified according to the location of metastasis (visceral [with or without bone metastases] vs. bone metastases alone) and PSA doubling time (≤ 3 vs. > 3 months). As per the standard of care, patients will have PSA testing performed every 6-12 weeks and re-imaging at 6, 9, 12, 18 and 24 months or at PSA progression, whichever occurs first.

The primary objective of this study will be to evaluate the radiographic progression-free survival. We also want to determine the time to the start of second line systemic therapy, the prostate-cancer specific survival, the overall survival as well as to assess the quality of life, the toxicity and the PSA response. This study is the first randomized study in this setting and will employ a randomized phase II design to determine if a larger scale phase III trial is needed, thus the phase II/III design. The Phase II will consist of 130 CRPC patients with oligometastases, and the phase III will consist of the already randomized 130 patients plus an estimated 244 patients for a total sample size of 374 patients. This study will be conducted through the Genitourinary Radiation Oncology Group of Quebec (GROUQ) in different radiation oncology centres across Canada and the recruitment should be completed within 30 months of activation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older and willing and able to provide informed consent;
2. Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features;
3. Ongoing androgen deprivation therapy with a Gonadotropin-releasing hormone (GnRH) analogue or bilateral orchiectomy (i.e., surgical or medical castration);
4. Patients who have not had a bilateral orchiectomy must have a plan to maintain effective GnRH analogue therapy for the duration of the trial;
5. Serum testosterone level ≤ 1.7 nmol/L (50 ng/dL) at the Screening visit;
6. Patients receiving bisphosphonate therapy/Xgeva must have been on stable doses for at least 4 weeks;
7. Progressive disease at study entry defined as one or more of the following three criteria that occurred while the patient was on androgen deprivation therapy as defined in eligibility criterion #3:

   1. PSA progression defined by a minimum of two rising PSA levels with an interval of ≥ 1 week between each determination. Patients who received an anti-androgen must have progression after withdrawal (≥ 4 weeks since last flutamide or ≥ 6 weeks since last bicalutamide or nilutamide). The PSA value at the Screening visit should be ≥ 2 μg/L (2 ng/mL);
   2. Metastatic disease documented by bone lesions on bone scan or by measurable soft tissue disease by CT/MRI. Patients whose disease spread is limited to regional pelvic lymph nodes, and previously radiated, are not eligible;

   i. Up to 5 metastatic sites ii. ≤ 4 tumours within any given organ system, excluding brain and liver (e.g. up to 4 bone metastases, or 4 lung metastases) iii. All sites of disease must be amenable to SBRT with no history of the metastases being irradiated; iv. In the case of a suspicious lesion in an unusual location such as lung or thoracic lymph nodes (without other abdominal lymph nodes), a biopsy should confirm prostate cancer origin.
8. No prior cytotoxic chemotherapy for prostate cancer;
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 or Karnofsky performance status of > 70% or higher;
10. Patients and their female partners of childbearing potential must be willing to use two forms of contraception (one of which must include a condom as a barrier method of contraception during sexual activity) throughout the duration of the study starting at screening and continuing for 3 months after the last dose of study drug or per local guidelines where these require additional description of birth control methods. These contraceptive methods must include the following:

    1. The use of condoms (barrier method)

       AND one of the following:
    2. the use of oral, injected or implanted hormonal methods of contraception by a female partner;
    3. placement of an intrauterine device (IUD) or intrauterine system (IUS) by a female partner;
    4. additional barrier method, such as occlusive cap (diaphragm or cervical/vault cap) with spermicidal foam/gel/film/cream/suppository by a female partner;
    5. tube ligation in the female partner;
    6. vasectomy or other procedure resulting in infertility (eg. bilateral orchiectomy) for ≥ 6 months.

    If the patient's partner is a pregnant woman, the patient must use a condom during sexual activity during and for 3 months after treatment with enzalutamide.
11. Patients must agree to not donate sperm while taking study drug
12. Estimated life expectancy of ≥ 6 months;
13. Ability to swallow the study drug whole and comply with study.

Exclusion Criteria:

1. Severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrollment;
2. Known or suspected brain metastasis or active leptomeningeal disease;
3. History of another malignancy within the previous 5 years other than curatively treated non-melanoma skin cancer;
4. Absolute neutrophil count < 1,500/μL, platelet count < 100,000/μL, or hemoglobin < 5.6 mmol/L (9 g/dL) at the Screening visit (NOTE: patients may not have received any growth factors within 7 days or blood transfusions within 28 days of the hematologic laboratory values obtained at the Screening visit);
5. Total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal at the Screening visit;
6. Creatinine > 177 μmol/L (2 mg/dL) at the Screening visit;
7. Albumin < 30 g/L (3.0 g/dL) at the Screening visit;
8. History of seizure or any condition that may predispose to seizure (e.g., prior cortical stroke or significant brain trauma). Also, history of loss of consciousness or transient ischemic attack within 12 months of enrollment (Day 1 visit);
9. Clinically significant cardiovascular disease including:

   1. Myocardial infarction within 6 months;
   2. Uncontrolled angina within 3 months;
   3. Congestive heart failure New York Heart Association (NYHA) class 3 or 4, or patients with history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multi-gated acquisition scan performed within three months results in a left ventricular ejection fraction that is ≥ 45%;
   4. History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes);
   5. History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place;
   6. Hypotension as indicated by systolic blood pressure < 86 millimeters of mercury (mmHg) at the Screening visit;
   7. Bradycardia as indicated by a heart rate of < 50 beats per minute on the Screening ECG;
   8. Uncontrolled hypertension as indicated by systolic blood pressure > 170 mmHg or diastolic blood pressure > 105 mmHg at the Screening visit.
10. Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within last 3 months);
11. Major surgery within 4 weeks of enrollment (Day 1 Visit);
12. Use of opiate analgesics (eg. morphine, fentanyl, etc.) for pain from prostate cancer within 4 weeks of enrollment (Day 1 visit). This does not apply to non-morphine drugs like codeine;
13. Radiation therapy for treatment of the primary tumour within 3 weeks of enrollment (Day 1 visit);
14. Radiation or radionuclide therapy for treatment of metastasis;
15. Primary disease not treated
16. More than 5 metastases
17. Hormone naïve prostate cancer patients
18. Treatment with flutamide within 4 weeks of enrollment (Day 1 visit);
19. Treatment with bicalutamide or nilutamide within 6 weeks of enrollment (Day 1 visit);
20. Treatment with 5-α reductase inhibitors (finasteride, dutasteride), estrogens, cytproterone within 4 weeks of enrollment (Day 1 visit)
21. Treatment with systemic biologic therapy for prostate cancer (other than approved bone targeted agents and GnRH-analogue therapy) or other agents with anti-tumour activity within 4 weeks of enrollment (Day 1 visit);
22. History of prostate cancer progression on ketoconazole;
23. Prior use, or participation in a clinical trial, of an investigational agent that blocks androgen synthesis (e.g., abiraterone acetate, TAK-700, TAK-683, TAK-448) or targets the androgen receptor (e.g., BMS 641988);
24. Participation in a previous clinical trial of enzalutamide;
25. Use of an investigational agent within 4 weeks of enrollment (Day 1 visit);
26. Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone per day within four weeks of enrollment (Day 1 visit);
27. Any condition or reason that, in the opinion of the Investigator, interferes with the ability of the patient to participate in the trial, which places the patient at undue risk, or complicates the interpretation of safety data.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2041-08 (Estimated)

PRIMARY OUTCOMES:
Radiographic Progression-free Survival | 5 years
  Time from randomization until disease progression confirmed by radiographic imaging or the start of new antineoplastic therapy.

SECONDARY OUTCOMES:
Quality of Life | 5 years
  Evaluate the impact of the treatment on the patient's quality of life using the FACT-P questionnaire
Quality of Life - Fatigue | 5 years
  Evaluate the impact of the treatment on the patient's quality of life using the Brief Fatigue Inventory (BFI) questionnaire
Quality of Life - Pain | 5 years
  Evaluate the impact of the treatment on the patient's quality of life using the Brief Pain Inventory (BPI) questionnaire
Toxicity | 5 years
  To determine acute and late toxicity due to radiotherapy, scored using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.3
Prostate Cancer Specific Survival | 5 years
  Time from randomization until death due to prostate cancer.
Time to Skeletal-related Event | 5 years
  Time from randomization until the occurrence of a skeletal related event (SRE).
Overall Survival | 5 years
  Time from randomization until death from any cause.
Local Control | 5 years
  To evaluate the impact of SBRT on oligometastases progression by radiographic imaging or the start of new antineoplastic therapy.
Time to Systemic Antineoplastic Therapy | 5 years
  Time from randomization to the administration of subsequent antineoplastic systemic therapy
PSA response | 5 years
  To evaluate PSA or the onset of biochemical failure
Predictive Value of Biomarkers | 5 years
  To evaluate the predictive value of the biomarkers in radiographic progression-free survival by analyzing for the presence or absence of biomarkers and evaluating for possible correlation with radiographic progression-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Tamim Niazi, MD, Principal Investigator — Jewish General Hospital
Locations (11):
- Canada (11):
  - BC CANCER Vancouver, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program - London Health Sciences Centre, London, Ontario
  - Hopital Charles-Lemoyne, Longueuil, Quebec
  - Centre Hospitalier de l'Université de Montréal (CHUM) - Hopital Notre Dame, Montreal, Quebec
  - Jewish General Hospital, McGill University, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - CHU de Quebec-Universite Laval, Québec, Quebec
  - Centre Hospitalier régional de Trois-Rivières, Trois-Rivières, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Niazi T, Saad F, Tisseverasinghe S, Koul R, Thibault I, Chung PWM, Wakil G, Lock M, Delouya G, Bahoric B, Feifer A, Agnihotram VR, Tsakiridis T, Cury FL, Dahmane R, Patil NG, Tyldesley S. Metastases-directed therapy in addition to standard systemic therapy in oligometastatic castration-resistant prostate cancer in Canada (GROUQ-PCS 9): a multicentre, open-label, randomised, phase 2 trial. Lancet Oncol. 2025 Sep;26(9):1158-1167. doi: 10.1016/S1470-2045(25)00351-1. PMID 40907514